CLINICAL TRIAL: NCT03379584
Title: A Phase 1 Study of SGN-CD48A in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Safety Study of SGN-CD48A in Patients With Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to overall benefit/risk profile
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGN48A-001
Record Dates: First submitted 2017-12-13; First posted 2017-12-20 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Antibody-drug conjugate
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SGN-CD48A (Experimental): SGN-CD48A
  Interventions: Drug: SGN-CD48A

INTERVENTIONS:
Drug: SGN-CD48A — Intravenous (IV) infusion on days 1, 8, and 15 of a 28-day cycle

SUMMARY:
This study will test the safety and activity of SGN-CD48A in patients with multiple myeloma. SGN-CD48A will be given on Days 1, 8, and 15 of a 28-day cycle. Prior to protocol amendment 2, SGN-CD48A was given every 3 weeks.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability, and antitumor activity of SGN-CD48A in patients with relapsed or refractory multiple myeloma. This study will be conducted in 2 parts:

1. Dose escalation: This part will evaluate increasing doses of SGN-CD48A to identify the maximum tolerated dose.

   The first group of patients enrolled on the study will receive the lowest dose of SGN-CD48A. Once this dose is shown to be safe, a second group of patients will be enrolled at the next higher dose. Patients will continue to be enrolled in groups receiving increasing doses until the maximum tolerated dose level is reached. Patients can only be enrolled into a higher dose level once the lower doses have been demonstrated safe. Dose escalation will be conducted using a modified toxicity probability interval (mTPI) study design.
2. Dose expansion: This part will further evaluate the safety, tolerability, and antitumor activity of up to 2 dose levels of SGN-CD48A shown to be safe in the first part of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MM requiring systemic therapy (per the International Myeloma Working Group [IMWG])
* Patients must not have other therapeutic options known to provide clinical benefit in MM available to them. Prior lines of therapy must include at least a proteasome inhibitor, an immunomodulatory drug, and an anti-CD38 antibody.
* Measureable disease, as defined by at least one of the following: serum M protein 0.5 g/dL or higher, urine M protein 200 mg/24 hour or higher, and serum immunoglobulin free light chain 10 mg/dL or higher and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Adequate hematologic, renal, and hepatic function
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy greater than 3 months
* A negative pregnancy test (for females of childbearing potential)
* Patients must provide written consent

Exclusion Criteria:

* Pre-existing peripheral neuropathy Grade 2 or higher
* History of malignancy other than MM within the past 3 years
* Active cerebral/meningeal disease related to the underlying malignancy
* Uncontrolled Grade 3 or higher infection
* Known to be positive for HIV or hepatitis B, or known to have active hepatitis C infection
* Previous allogeneic stem cell transplant
* History of cerebral vascular event, unstable angina, myocardial infarction, or cardiac symptoms consistent with congestive heart failure within the last 6 months
* Treatment with any known P-gp inducers/inhibitors or strong CYP3A inhibitors within 14 days prior to the first dose of study drug
* Prior antitumor therapy that is not completed at least 4 weeks prior to first dose of study drug, or at least 2 weeks if progressing. Prior CAR T-cell therapy must be completed 8 weeks before first dose of study drug.
* Females who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Type, incidence, severity, seriousness, and relatedness of adverse events | Through 1 month following last dose
Incidence of laboratory abnormalities | Through 1 month following last dose
Incidence of dose limiting toxicity | Through 3 weeks following first dose

SECONDARY OUTCOMES:
Objective response rate | Through 1 month following last dose
  The proportion of patients with stringent complete response, complete response, very good partial response, or partial response per investigator
Complete response rate | Through 1 month following last dose
  The proportion of patients with stringent complete response or complete response per investigator
Duration of objective response | Up to approximately 3 years
Duration of complete response | Up to approximately 3 years
Progression-free survival | Up to approximately 3 years
Overall survival | Up to approximately 3 years
Blood concentrations of SGN-CD48A and metabolites | Through 1 month following last dose
Incidence of antitherapeutic antibodies | Through 1 month following last dose

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne McGoldrick, MD, MPH, Study Director — Seagen Inc.
Locations (6):
- United States (6):
  - University of California at San Francisco, San Francisco, California
  - Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Mount Sinai Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania / Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania